CLINICAL TRIAL: NCT05978921
Title: Effect of Physical Strength Exercise on Telomeric Length as a Marker of Aging and Early Death in Patients With Schizophrenia
Brief Title: Physical Exercise in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Juan Luis Sanchez Gonzalez, Principal Investigator. Juan Luis Sánchez González, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ExerciseSchizophrenia
Record Dates: First submitted 2023-07-17; First posted 2023-08-07 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Schizophrenia; Physical Activity; Telomere Shortening; Premature Aging
MeSH Terms: conditions — Schizophrenia; Motor Activity; Aging, Premature

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The persons in charge of the evaluation of the participants will be unaware of the assignment of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): An additional strength training programme will be carried out for 12 weeks with 2 sessions per week. The sessions will last approximately 50 minutes and will be divided into 3 distinct parts: The first part will consist of a warm-up with a part of aerobic exercise that will last approximately 15 minutes. This will be followed by the main part of strength training with a circuit of 6 exercises (3 series x 12 repetitions) which will last approximately 25 minutes.
  Finally, there will be a cool down phase with breathing exercises to allow people to recover.
  Interventions: Other: Strength physical exercise programme
- Control group (Sham Comparator): Subjects in the control group will continue with their normal life and carry out all the activities they have been doing previously.
  Interventions: Other: Normal life

INTERVENTIONS:
Other: Strength physical exercise programme — 12 multi-joint strength exercises will be developed. Participants will be taught the rating scale of perceived exertion (RPE) based on the number of repetitions in reserve (RIR). Participants will be asked that during the performance of each of the exercises they must perceive an effort between 7-8 within the overall score of the scale (0-10; 0 = no effort at all and 10 = cannot perform one more repetition, i.e. maximal effort). When subjects perform the 12 repetitions with lower perceived exertion than the set effort in two consecutive sessions with full range of motion the training load will be increased by about 2-10% following the American College of Sports Medicine guidelines and reassessed using the RIR-based RPE. Patients in the usual treatment group will continue to participate in their existing rehabilitation programmes, but will not be included in the strength training programme.
  Arms: Intervention group
Other: Normal life — Normal life and carry out all the activities they have been doing previously.
  Arms: Control group

SUMMARY:
Randomised clinical trial on a cohort of subjects with a diagnosis of schizophrenia of legal age, of both sexes, recruited in the mental health clinics of the Salamanca University Assistance Complex and who will be randomly distributed into two groups (intervention and control).

The main objective of the study is to determine the effect of physical exercise on telomere size in patients diagnosed with schizophrenia.

As secondary objectives in this group of patients we will try to:

Evaluate the influence of strength training on cognition and negative symptoms of schizophrenia.

To quantify the impact of strength training on frailty. To determine the effect of strength training on quality of life. To study the possible correlation between physical parameters (frailty) and telomere length.

To establish the importance of polymorphisms in telomerase genes, an enzyme involved in the maintenance of telomere length.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* have been diagnosed with schizophrenia for at least 5 years

Exclusion Criteria:

* are unable to read and understand the patient information sheet and sign the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Telomere Length | Baseline and immediately after the intervention
  Telomere length will be measured before and after the procedure in kilobases.

SECONDARY OUTCOMES:
Date of birth | Baseline
  It will be registered at the beginning of the study in order to calculate the age of the participant.
Sex | Baseline
  It will be registered at the beginning of the study.
Heighth | Baseline
  It will be registered at the beginning of the study in centimeters.
Negative Symptoms | Baseline and immediately after the intervention
  Negative symptoms of the disease will be measured and assessed using the Brief Negative Symptom Scale (BNSS). The BNSS is comprised of 13 questions organized into 6 subscales that assess anhedonia, distress, asociality, avolition, blunted affect, and alogia. Items are scored on a 0 to 6 scale, with 0 indicating the symptom is absent and 6 indicating the symptom is severe
Fragility | Baseline and immediately after the intervention
  Fragility will be measured using the Short Physical Performance Battery scale (SPPB). SPPB scores range from zero to 12 possible points. SPPB score of 3-9 points in persons with possible sarcopenia but no mobility disability indicates frailty; SPPB score of 10 or greater for persons with no sarcopenia and no mobility disability indicates robustness. Persons with a score of 2 or lower who have sarcopenia, potential cachexia, and mobility disability are determined to be disabled.
Cognition | Baseline and immediately after the intervention
  Cognition will be measured using the Brief Assessment of Cognition in Schizophrenia (BACS).The maximum and minimum score on the Brief Assessment of Cognition in Schizophrenia (BACS) is 100 points and the minimum possible score is 0 points. The scoring scale is based on the performance of a normative reference group, where the mean is set at 100 and the standard deviation at 15. Thus, a score of 100 indicates average performance within the normative population, while a higher score would be considered above average and a lower score below average.
Quality of life | Baseline and immediately after the intervention
  Quality of life will be assessed using the EuroQuality of Life (EQ-5D-5L scale). This scale is numbered from 0 to 100. • 100 means the best health you can imagine. 0 means the worst health you can imagine.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Castilla Y León / Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Upon request by e-mail to the principal investigator